CLINICAL TRIAL: NCT04580927
Title: Improving Cardiovascular Health in New Mothers: Multi-Centre Open-Label Randomized Trial of a Breastfeeding Intervention to Improve Breastfeeding Practices and Lower Blood Pressure in Women With Hypertensive Disorders of Pregnancy
Brief Title: Breastfeeding and Postpartum Cardiovascular Health
Acronym: sheMATTERS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); McGill University (Other)
Responsible Party: Principal Investigator, Natalie Dayan, Physician and Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MP-37-2021-7201: she MATTERS
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Hypertensive Disorder of Pregnancy; Pregnancy Complications; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Breastfeeding
MeSH Terms: conditions — Toxemia; Pregnancy Complications; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Multi-site open-label, randomized control trial, evaluating a nurse-led breastfeeding self-efficacy enhancing intervention for women who had hypertensive disorders of pregnancy recruited at three sites in Canada. Participants that plan to breastfeed will be randomly divided into two groups: one will be given the BSE intervention, the other will not. Both groups will receive same standard postpartum care: routine postpartum hospital breastfeeding support, community breastfeeding support, and postpartum medical visits with obstetrics care provider and cardiovascular risk assessment. Participants who had high blood pressure in pregnancy and are not planning to breastfeed will not be randomized and will receive standard postpartum care excluding breastfeeding care. Outcomes for all participants will be assessed by completion of questionnaires, collecting blood pressure measurements and blood tests and long-term follow-up via linkage with administrative health data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomized to breastfeeding self-efficacy enhancing intervention with nurse (Experimental): Participants receiving breastfeeding self-efficacy enhancing nurse-led intervention plus postpartum standard of care consisting of postpartum medical visits with their obstetrics care provider and for cardiovascular risk assessment, routine postpartum hospital breastfeeding support, as-needed community breastfeeding support, and postpartum medical visits with their obstetrics care provider and for cardiovascular risk assessment.
  Interventions: Behavioral: Breastfeeding self-efficacy (BSE)
- Randomized to usual postpartum care (No Intervention): Participants receiving postpartum standard of care consisting of postpartum medical visits with their obstetrics care provider and for cardiovascular risk assessment, routine postpartum hospital breastfeeding support, as-needed community breastfeeding support, and postpartum medical visits with their obstetrics care provider and for cardiovascular risk assessment.
- Non-randomized observational arm (No Intervention): Participants who are not planning to breastfeed receiving postpartum standard of care consisting of postpartum medical visits with their obstetrics care provider and for cardiovascular risk assessment.

INTERVENTIONS:
Behavioral: Breastfeeding self-efficacy (BSE) — Self-efficacy is determined by factors such as prior experience, vicarious learning, persuasion of others and physiological state, which in turn impact on one's behaviours and actions. One's sense of self-efficacy is modifiable, and can be readily targeted for intervention. An increasingly studied key determinant of breastfeeding outcomes is breastfeeding confidence, also referred to as breastfeeding self-efficacy (BSE). The investigators will use a nurse-administered validated BSE intervention tool.
  Arms: Randomized to breastfeeding self-efficacy enhancing intervention with nurse

SUMMARY:
Hypertensive disorders of pregnancy (HDP) are increasingly recognized sex-specific risk factors for premature cardiovascular disease (CVD) in women. HDP, including preeclampsia and gestational hypertension, confer a 2- to 3-fold increase in the risk of chronic hypertension and ischemic heart disease 10-15 years after delivery. Observational data suggest that breastfeeding can lower maternal blood pressure (BP), risk of metabolic syndrome, and other markers of cardiovascular risk in the short term and long term, possibly by helping to re-set the metabolic changes of pregnancy. The investigators recently demonstrated an 11% reduction in the risk of metabolic syndrome among postpartum women with a variety of complications in pregnancy, including HDP, who breastfed for > 6 months, compared to those who did not breastfeed and those who breastfed for shorter durations. An analysis of 622 postpartum women at Kingston General Hospital showed that breastfeeding women had nearly a 6-mmHg lower systolic BP than women who did not breastfeed with an apparent dose-response effect of breastfeeding duration. Women with pregnancy complications including HDP are vulnerable to early weaning. Interactive, multi-modal approaches targeting a mother's breastfeeding self-efficacy (i.e., confidence about breastfeeding) have been effective in healthy postpartum women. However, these have not yet been tested specifically in HDP women, who stand to derive substantial benefit from breastfeeding. This is an important area to study since nurse-led breastfeeding supportive interventions can be widely applied to the postpartum care of women with HDP and can be integrated into comprehensive CVD risk reduction programs for these women. The primary outcome is postpartum BP, since hypertension is a key mediating factor in women's heart health. The investigators conducted a feasibility study of a breastfeeding self-efficacy intervention to enhance breastfeeding outcomes among women with HDP achieving pre-defined targets of a recruitment rate of >50% , attrition rates of < 30%, and > 70% participant satisfaction with the intervention, measured at the 6-month time point. Additionally, data showed trends in both systolic and diastolic BP favoring the intervention group. The current study is a multi-site open-label randomized trial to assess for a difference in blood pressure and breastfeeding between groups, and to serve as a cohort of HDP women for longitudinal follow-up.

DETAILED DESCRIPTION:
The present study aims to assess a nurse-led self-efficacy enhancing breastfeeding intervention in women who have HDP. The investigators will examine whether this intervention reduces postpartum blood pressure and improves breastfeeding outcomes in these women. In the long-term, the investigators will observe to see whether breastfeeding helps to lower the chance of chronic hypertension or other cardiovascular risk factors, as well as heart disease or stroke.

Outcomes:

As per study protocol amendment approved by the RI-MUHC Research Ethics Board on July 2023, all study aims (with the exception of the exploratory ones such as Objective 8, Biomarkers) now address an active 6-months follow up period, and a passive 12-months follow up allowing a shorter time for data analysis and study completion. This modification will align the end of study with the availability of funding resources.

Previously, it was stated that "All outcomes will be ascertained at the end of the study, which is at 12 months postpartum."

The primary study endpoint is systolic and/or diastolic BP, in mmHg.

Secondary study endpoints:

* Breastfeeding outcomes: i. Duration of exclusive breastfeeding (weeks); ii. The proportion who breastfeed (exclusive or non-exclusive) at 6 months;
* The presence of metabolic syndrome.

Additional objectives:

-to evaluate whether women who breastfeed for longer are more likely to engage in cardiovascular protective behaviors such as weight reduction, healthy eating and higher levels of physical activity at 12 months postpartum; to explore the biological and psychosocial determinants of breastfeeding behaviour within 12 months postpartum, measured at the time of delivery; to assess the risk of future hospitalization or emergency room visit for any cardiovascular event or procedure within 15 years after delivery, according to: (a) breastfeeding intervention, (b) total duration of breastfeeding, and (c) other novel determinants of cardiovascular risk; to collect biosamples among women who recently had HDP, in order to advance on the understanding of the different phenotypes of women and their associated cardio-metabolic risk in the short and long-term.

Women who had HDP will be recruited from three participating centers. In Quebec there will be three (previously two) centers: (1) McGill University Health Centre-Royal Victoria Hospital (MUHC-RVH) and (2) St. Mary's Hospital Centre (SMHC) and the Jewish General Hospital (JGH), the fourth (previously third) site will be in Ontario at the (3) Kingston General Hospital (KGH). Participants that plan to breastfeed will be randomly divided into two groups: usual postpartum care + BSE intervention or usual postpartum care. Participants with HDP who are not planning to breastfeed will also be invited to participate as an additional observational comparison group. Study outcomes for all participants will be assessed by completion of questionnaires, home and in-office blood pressure measurement, basic metabolic biochemical testing and long-term follow-up via linkage with administrative health data.

NOTE: The pandemic and other factors have led to delays in approvals at different sites, and associated challenges with recruitment. Due to these delays and funding deadlines, we revised sample size calculation with more realistic and less stringent assumptions. Sample size was modified from 323 to 221. This modification was approved by the RI-MUHC Research Ethics Board on July 2023

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Singleton live birth delivered at >34 weeks gestation.
* Mother intends to breastfeed (randomized portion)
* Breastfeeding initiated before postpartum hospital discharge (randomized portion)
* Participant speaks and understands English or French.
* Participant has a valid Medicare card (RAMQ, OHIP) at time of recruitment.
* Participant has access to a cellular telephone to receive text messages and install a Blood Pressure Monitoring Application, and internet access to receive emails and to complete online questionnaires.
* Be available to attend in-person visits if COVID restrictions allow (resides in Montreal, Kingston or surrounding areas)
* Have AT LEAST ONE OR MORE of the criteria listed below related to the diagnosis of HDP:

  i. Pregnancy at or beyond 20 weeks gestation with: Two (2) recorded seated BPs taken at least 15 minutes apart during one medical visit measuring >140 mmHg systolic AND/OR >90 mmHg diastolic AND Recorded elevated BP is present at more than one consecutive medical visit ii. Women who during antenatal visits were prescribed antihypertensive medication, OR received a diagnosis of chronic or gestational hypertension iii. Women who during labor and delivery, had two (2) or more BP measurements >140 mmHg systolic or >90 mmHg diastolic at least 15 minutes apart or who were prescribed antihypertensive medication iv. Women who during labor and delivery received a diagnosis of preeclampsia v. Women with new-onset hypertension as defined above, and/or preeclampsia and/or pre-existing hypertension readmitted within 1 week of postnatal hospital discharge with elevated blood pressure.

Exclusion Criteria:

Exclusion criteria from randomized trial portion of the study:

* Maternal absolute contraindication to breastfeeding (e.g., mother taking medication for which breastfeeding is contraindicated , or mother is infected with human immunodeficiency virus, HTLV-1, active tuberculosis, active herpes simplex on the breast, or Ebola, or mother is a cocaine or phencyclidine user).
* Maternal condition that interferes with breastfeeding (e.g., breast reduction, or breast augmentation surgery due to hypoplastic mammary tissue. Uncomplicated breast augmentation surgery is not an exclusion criterion).
* Neonatal absolute contraindication to breastfeeding (Galactosemia)
* Neonatal condition that interferes with breastfeeding (e.g., cleft palate).

Exclusion criteria from randomized OR observational portion of the study (including non-randomized arm):

* Infant born before 34 weeks gestation.
* Maternal intensive care unit (ICU) admission lasting >24 hours.
* Severe or uncontrolled psychiatric illness in the mother that would preclude active engagement in the study. These include schizophrenia or other psychotic disorder; uncontrolled bipolar disorder; major depressive episode within the last year, or history of major depressive disorder requiring hospitalization at any point; substance abuse disorder; any previous suicide attempt.
* Mother has active COVID-19 infection (confirmed by positive COVID test) at time of postpartum hospitalization.
* Previous BP-MOM participant (ISRCTN85493925, www.isrctn.com)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who had high blood pressure in pregnancy
Enrollment: 221 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Lower Systolic and/or diastolic BP, in mmHg. | 6 months and passive follow up until 12 months
  Evaluate whether a nurse-led BSE intervention will result in a lower systolic and/or diastolic BP 6 months (and passive follow up to 12 months) postpartum
Number of Participants Using Antihypertensive Therapy | 6 months and passive follow up until 12 months
  Evaluate whether a nurse-led BSE intervention will result in a lower need for antihypertensive therapy

SECONDARY OUTCOMES:
Number of Participants Providing Exclusive Breastfeeding (weeks) | 6 months and passive follow up until 12 months
  Evaluate whether a nurse-led BSE intervention will result in longer duration of exclusive breastfeeding
Proportion of Participants who Breastfeed (exclusive or non-exclusive) | 6 months and passive follow up until 12 months
  Evaluate whether a nurse-led BSE intervention will result in higher rates of any continued breastfeeding at 6 months
Number of Participants that Develop Metabolic Syndrome | 6 months and passive follow up until 12 months
  Evaluate whether a nurse-led BSE intervention will result in lower metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Dayan, MD, MSc, Study Director — McGill University Health Center- Research Institute of the McGill University Health Center; Sonia Semenic, N, PhD, Principal Investigator — Associate Professor and PhD Program Ingram School of Nursing, McGill University; Graeme Smith, MD, PhD, Principal Investigator — Prof. Head Dept Obstetrics - Gynaecology, Dept. Biomedical and Molecular Sciences Queen's University; Atanas Nedelchev, MD, Principal Investigator — Assistant Professor, Department of Obstetrics and Gynecology; Haim Abenhaim, MD, MPH, Principal Investigator — Jewish General Hospital
Locations (4):
- Canada (4):
  - Kingston General Hospital, Kingston, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - St Mary's Hospital, Montreal, Quebec
  - Muhc-Rimuhc, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
The plan to share is not defined yet

REFERENCES:
- [Result] Yu J, Pudwell J, Dayan N, Smith GN. Postpartum Breastfeeding and Cardiovascular Risk Assessment in Women Following Pregnancy Complications. J Womens Health (Larchmt). 2020 May;29(5):627-635. doi: 10.1089/jwh.2019.7894. Epub 2019 Dec 3. PMID 31800357
- [Result] Smith GN, Pudwell J, Roddy M. The Maternal Health Clinic: a new window of opportunity for early heart disease risk screening and intervention for women with pregnancy complications. J Obstet Gynaecol Can. 2013 Sep;35(9):831-839. doi: 10.1016/S1701-2163(15)30841-0. No abstract available. PMID 24099450
- [Result] Dennis CL. Theoretical underpinnings of breastfeeding confidence: a self-efficacy framework. J Hum Lact. 1999 Sep;15(3):195-201. doi: 10.1177/089033449901500303. No abstract available. PMID 10578797
- [Result] Dennis CL, McQueen K. The relationship between infant-feeding outcomes and postpartum depression: a qualitative systematic review. Pediatrics. 2009 Apr;123(4):e736-51. doi: 10.1542/peds.2008-1629. PMID 19336362
- [Result] Grand'Maison S, Pilote L, Okano M, Landry T, Dayan N. Markers of Vascular Dysfunction After Hypertensive Disorders of Pregnancy: A Systematic Review and Meta-Analysis. Hypertension. 2016 Dec;68(6):1447-1458. doi: 10.1161/HYPERTENSIONAHA.116.07907. Epub 2016 Oct 17. PMID 27754864
- [Derived] Dayan N, Smith G, Nedelchev A, Abenhaim H, Brown R, Da Costa D, Ali S, Perlman J, Nguyen TV, Dennis CL, Abdelmageed W, Semenic S. Study protocol for the sheMATTERS study (iMproving cArdiovascular healTh in new moThERS): a randomized behavioral trial assessing the effect of a self-efficacy enhancing breastfeeding intervention on postpartum blood pressure and breastfeeding continuation in women with hypertensive disorders of pregnancy. BMC Pregnancy Childbirth. 2023 Jan 26;23(1):68. doi: 10.1186/s12884-022-05325-3. PMID 36703104